CLINICAL TRIAL: NCT00773656
Title: Surveillance of the Cohort of Patients Overexposed in a Course of Conformational Radiotherapy for a Prostate Adenocarcinoma in Jean MONNET Hospital, Epinal, France. Epinal: Patients Overexposed for a Prostate Adenocarcinoma
Brief Title: Patients Overexposed for a Prostate Adenocarcinoma
Acronym: EPOPA
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: AOM 08234
Record Dates: First submitted 2008-10-15; First posted 2008-10-16 (Estimated); Last update posted 2014-02-27 (Estimated); Status verified 2014-02

CONDITIONS: Prostate Adenocarcinoma
Keywords: Radiotherapy; Biologically effective dose; Radiation injury
MeSH Terms: conditions — Radiation Injuries

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — White cells, serum and DNA
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- 1: patients treated for a prostate adenocarcinoma
  Interventions: Other: Whole blood sample

INTERVENTIONS:
Other: Whole blood sample — 70 ml per patient for collection of biological sample

SUMMARY:
Background:

Between 2000 and 2006, 433 patients were overexposed (8% to 10%) during a course of conformal radiotherapy for a prostate adenocarcinoma in Jean MONNET hospital, Epinal, France. Among them, twenty four patients received an additional mean dose about 20%, due to an inappropriate use of the treatment planning system. Severe adverse events (proctitis, cystitis, and tissue necrosis) have occurred among most of these overexposed patients. We propose to develop several research programs in order to increase the scientific knowledge on iatrogenic effects related to overexposure of ionizing radiation, by studying their relationship with dosimetric, clinical, biologic and genetic characteristics.

Aim of the study:

To correlate the received doses, the volume of irradiated normal tissues, the events, with biologic, phenotypic and genetic data.

Primary study endpoint:

Incidence and severity of adverse events related to radiotherapy (according to SOMA - LENT and CTCAE scales).

DETAILED DESCRIPTION:
Secondary study endpoint:

* Correlation between adverse events and radiation doses with biologic, phenotypic and genetic data.
* Evaluation of T-lymphocyte apoptosis to predict radiation-induced late toxicity
* Gene associations with risks for adverse events related to radiotherapy
* Levels of circulating microparticles and bystander effect after irradiation

Inclusion criteria:

Consecutive patients treated for a prostate adenocarcinoma in the radiation department of the Jean MONNET Hospital between 2000 and 2006.

Potential. Better identification of patients at high risk of adverse events related to radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* provision of informed consent
* patient treated for prostate adenocarcinoma and overexposed during radiotherapy in a prostate adenocarcinoma in the radiation department of the a prostate adenocarcinoma in the radiation department of the Jean MONNET hospital/ service de radiotherapies between 2000 and 2006

Exclusion Criteria:

* No provision of informed consent
* Patient with disease worsening and in incapacity to move about to CHJM

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients treated for a prostate adenocarcinoma in the radiation department of the Jean MONNET Hospital between 2000 and 2006.
Sampling Method: Non-Probability Sample
Enrollment: 249 (Actual)
Dates: Start 2008-10; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
To correlate the received doses, the volume of irradiated normal tissues, the events, with biologic, phenotypic and genetic data. | At the inclusion visit

SECONDARY OUTCOMES:
Correlation between adverse events and radiation doses with biologic, phenotypic and genetic data. | At the inclusion visit
Evaluation of T-lymphocyte apoptosis to predict radiation-induced late toxicity | At the inclusion visit
Gene associations with risks for adverse events related to radiotherapy | At the inclusion visit
Levels of circulating microparticles and bystander effect after irradiation | At the inclusion visit

CONTACTS AND LOCATIONS:
Overall Officials: Jean Marc SIMON, PH, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Groupe Hospitalier Pitié-Salpêtrière, Paris, France

REFERENCES:
- [Background] Alsbeih G, El-Sebaie M, Al-Harbi N, Al-Buhairi M, Al-Hadyan K, Al-Rajhi N. Radiosensitivity of human fibroblasts is associated with amino acid substitution variants in susceptible genes and correlates with the number of risk alleles. Int J Radiat Oncol Biol Phys. 2007 May 1;68(1):229-35. doi: 10.1016/j.ijrobp.2006.12.050. Epub 2007 Feb 27. PMID 17331670
- [Derived] Ribault A, Benadjaoud MA, Squiban C, Arnaud L, Judicone C, Leroyer AS, Rousseau A, Huet C, Guha C, Benderitter M, Lacroix R, Flamant S, Chen EI, Simon JM, Tamarat R. Circulating microvesicles correlate with radiation proctitis complication after radiotherapy. Sci Rep. 2023 Feb 4;13(1):2033. doi: 10.1038/s41598-022-21726-y. PMID 36739457